CLINICAL TRIAL: NCT07306325
Title: Effectiveness of Ultrasonography in Evaluating the Airway and Predicting Difficult Intubation in Patients Diagnosed With Acromegaly
Brief Title: Ultrasound in Predicting Difficult Intubation in Acromegaly Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Muzaffer GENCER, Associate Professor Doctor, Başakşehir Çam & Sakura City Hospital
Other Study IDs: BSH-RG-Difficult Intubation
Record Dates: First submitted 2024-11-24; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Acromegaly Due to Pituitary Adenoma; Difficult Intubation; Airway Ultrasonography
Keywords: difficult intubation; acromegaly; airway ultrasonography
MeSH Terms: conditions — Growth Hormone-Secreting Pituitary Adenoma; Acromegaly | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants diagnosed with acromegaly: All ultrasonographic assessments will be performed preoperatively by anesthesiologists who have prior experience using ultrasound. Participants will be positioned in the supine position with the head and neck in neutral alignment. Measurements of the skin-hyoid bone, skin-epiglottis, and skin-anterior commissure of the vocal cords distances will be.
  Endotracheal intubation of the participants will be performed by anesthesiologists who are unfamiliar with the ultrasonographic measurements. During the intubation, the use of adjuncts, the need for cricoid pressure, the number of additional interventions, the number of additional operators, and the glottic opening seen during laryngoscopy will be recorded according to the Cormack-Lehane classification without external pressure. If necessary, advanced airway devices (videolaryngoscopy, flexible fiberoptic laryngoscopy) will be used.
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — In participants diagnosed with acromegaly, every patient to whom USG measurement methods are applied is followed by researchers before, during and after anesthesia applications, whether or not they are included in any study . Routine treatments that participants need will be fully implemented. Preoperative, intraoperative and postoperative follow-up data, which will be recorded observationally, will be used in this study.

SUMMARY:
This is a prospective observational study.The purpose of this study is to predict difficult intubation with ultrasonographic evaluation combined with preoperative physical examination in patients diagnosed with acromegaly and planned for pituitary surgery.

DETAILED DESCRIPTION:
Airway management is an important issue for patient safety in anesthesia. Difficult ventilation and difficult intubation are important causes of anesthesia-related perioperative morbidity and mortality. It is reported that approximately 30% of anesthesia-related mortality is related to inadequacy in difficult airway management. The incidence of difficult intubation is 1.5-13.2% in the general population.

Features evaluated for difficult airway risk prediction: age, gender, body mass index, weight, height, history of difficult intubation, facial and jaw features, mouth opening, head and neck mobility, prominent upper incisors, presence of beard, upper lip bite test, mallampati score, thyromental distance, hyomental distance , sternomental distance includes the distance between the incisors.

Acromegaly is an endocrinological disease with significant mortality and morbidity due to high growth hormone (GH) and insulin-like growth factor-I (IGF-I) levels. It usually occurs due to a pituitary tumor. Excessive GH secretion in adults causes acromegaly with overgrowth in the acral areas. Acral changes seen in these patients may cause abnormal airway structure and, accordingly, airway management may become difficult during anesthesia. Typically, large nose and tongue, thick mandible, and thick and large lips can be observed in acromegaly. There is hypertrophy in the pharynx, larynx, tonsil, vocal cords, mucosa and soft tissues. These features of acromegaly may cause difficult mask ventilation and difficult intubation. The incidence of difficult intubation is observed to be 10%-30% in acromegalic individuals.

With developing technology, the use of ultrasonography in preoperative airway evaluation has become widespread. It is a real-time, non-invasive, easily accessible, mobile, safe, painless method that can be used to evaluate both the upper and lower airway. Clinical airway screening tests aim to predict difficult airways. Recent reviews have shown that ultrasonographic measurements have a greater predictive value than airway screening tests performed by physical examination. Measurements obtained from ultrasound include skin-vocal cord distance, skin-hyoid distance and skin-epiglotte distance.

In the preoperative physical examination; Age, gender, height, weight, body mass index, mouth opening, neck extension, mallampati score, thyromental-hyomental and sternomental distance, neck circumference measurement and upper lip bite test will be evaluated.

All airway ultrasonographic evaluations will be performed preoperatively by experienced anesthesiologists who have previously performed airway ultrasonography. Participants will be prepared for ultrasonographic evaluation in the supine position, and skin-hyoid bone, skin-epiglotte, skin-vocal cord anterior commissure distance measurements will be made and recorded.

Intubation of the participants will be performed by experienced anesthesiologists who are unfamiliar with ultrasonography measurements.The assistive stylet used during the intubation of the participants, the need for cricoid pressure, the number of attempts, the number of practitioners and the glottis opening seen during laryngoscopy will be noted in accordance with the Cormack Lehane classification.Advanced airway devices will be used when necessary.

Preoperative physical examination values, ultrasonographic measurements and blood test results of the participants will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* • Patients diagnosed with acromegaly who are planned for endoscopic pituitary surgery

  * Volunteer participants
  * American Society of Anesthesiology - ASA 1, 2 and 3 patient groups
  * Patients with BMI<40

Exclusion Criteria:

* ASA 4 patient group

  * History of previous neck surgery
  * Patients with a history of tracheostomy
  * Patients with a history of radiotherapy to the neck area
  * Patients with limited neck extension (rheumatological - traumatic reasons)
  * Patients with masses and lesions in the mouth and airway that may make intubation difficult.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-70, regardless of gender, who are scheduled for endoscopic pituitary surgery at Başakşehir Çam and Sakura City Hospital Neurosurgery Clinic, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Airway Ultrasonography | one year
  Sonoatomonic evaluation of the airway and determination of difficult intubation in participants diagnosed with acromegaly and planned for pituitary surgery. - Distance Between Skin-Hyoid Bone (centimeters):
Airway Ultrasonography | one year
  Sonoatomonic evaluation of the airway and determination of difficult intubation in participants diagnosed with acromegaly and planned for pituitary surgery. - Distance Between Skin-Epiglottis (centimeters):
Airway Ultrasonography | one year
  Sonoatomonic evaluation of the airway and determination of difficult intubation in participants diagnosed with acromegaly and planned for pituitary surgery. - Distance Between Skin-Vocal Cord Anterior Commissure (centimeters)

SECONDARY OUTCOMES:
preoperative physical examination | one year
  Prediction of difficult intubation in participants diagnosed with acromegaly using classical airway examination tests
  -Age(year)
preoperative physical examination | one year
  Prediction of difficult intubation in participants diagnosed with acromegaly using classical airway examination tests
  -Gender:
preoperative physical examination | one year
  Prediction of difficult intubation in participants diagnosed with acromegaly using classical airway examination tests -Height(centimeters)
preoperative physical examination | one year
  Prediction of difficult intubation in participants diagnosed with acromegaly using classical airway examination tests
  * weight(kilograms)
preoperative physical examination | one year
  Prediction of difficult intubation in participants diagnosed with acromegaly using classical airway examination tests
  * BMI(kg/m^2):
preoperative physical examination | one year
  Prediction of difficult intubation in participants diagnosed with acromegaly using classical airway examination tests -Thyromental Distance(centimeters)
preoperative physical examination | one year
  Prediction of difficult intubation in participants diagnosed with acromegaly using classical airway examination tests -Stenomental Distance(centimeters) :
preoperative physical examination | one year
  Prediction of difficult intubation in participants diagnosed with acromegaly using classical airway examination tests - Upper Lip Biting Test:
preoperative physical examination | one year
  Prediction of difficult intubation in participants diagnosed with acromegaly using classical airway examination tests - Mallampati Score:
correlation with laboratory | one year
  Does difficult intubation become more frequent as growth hormone levels (nanograms/milliliter) increase?
correlation with laboratory | one year
  Does difficult intubation become more frequent as insulin-like growth hormone- 1 levels (micrograms/liter) increase?

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam ve Sakura Hastanesi, Istanbul, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Apfelbaum JL, Hagberg CA, Connis RT, Abdelmalak BB, Agarkar M, Dutton RP, Fiadjoe JE, Greif R, Klock PA, Mercier D, Myatra SN, O'Sullivan EP, Rosenblatt WH, Sorbello M, Tung A. 2022 American Society of Anesthesiologists Practice Guidelines for Management of the Difficult Airway. Anesthesiology. 2022 Jan 1;136(1):31-81. doi: 10.1097/ALN.0000000000004002. PMID 34762729
- [Background] Kasinath MPR, Rastogi A, Priya V, Singh TK, Mishra P, Pant KC. Comparison of Airway Ultrasound Indices and Clinical Assessment for the Prediction of Difficult Laryngoscopy in Elective Surgical Patients: A Prospective Observational Study. Anesth Essays Res. 2021 Jan-Mar;15(1):51-56. doi: 10.4103/aer.aer_75_21. Epub 2021 Aug 30. PMID 34667348
- [Background] Rao S, Paliwal N, Saharan S, Bihani P, Jaju R, Sharma UD, Sharma M. A Comparative Study to Evaluate Difficult Intubation Using Ratio of Patient Height to Thyromental Distance, Ratio of Neck Circumference to Thyromental Distance and Thyromental Height in Adult Patients in Tertiary Care Centre. Turk J Anaesthesiol Reanim. 2023 Apr;51(2):90-96. doi: 10.5152/TJAR.2022.22077. PMID 37140573
- See also: Related Info — https://jag.journalagent.com/z4/vi.asp?pdir=anestezi&plng=tur&un=JARSS-00710